CLINICAL TRIAL: NCT01622023
Title: Timing of IUI 24 or 48 Hours After Spontaneous LH Peak: a Randomised Controlled Trial
Brief Title: Timing of Intrauterine Insemination (IUI) 24 or 48 Hours After Spontaneous Luteinizing Hormone (LH) Peak
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Blockeel Christophe, MD, PhD, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1/2012
Record Dates: First submitted 2012-03-27; First posted 2012-06-18 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Pregnancy
Keywords: insemination; donor sperm; natural cycle

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study group (Experimental): intrauterine insemination after 24 hours
  Interventions: Procedure: intra-uterine insemination
- Control group (Active Comparator): intrauterine insemination after 48 hours
  Interventions: Procedure: intra-uterine insemination

INTERVENTIONS:
Procedure: intra-uterine insemination — Artificial insemination is the process by which sperm is placed into the reproductive tract of a female for the purpose of impregnating the female by using means other than sexual intercourse or natural insemination.
  Other Names: no other interventions

SUMMARY:
The aim of the present study is to prospectively evaluate whether performing an intra-uterine insemination 24 hours after the spontaneous LH peak may result in significantly higher ongoing pregnancy rates compared to 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* below 39 years of age on the day of LH peak
* donor semen
* natural cycle (without CC)
* cycle with less than 3 follicles reaching 15 mm of diameter or more.
* with basal hormonal values of progesterone ( < 1,2 ng/dl)

Exclusion Criteria:

The patients excluded are women

* who underwent more than 6 intrauterine inseminations,
* with tubal infertility

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 435 (Actual)
Dates: Start 2010-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
pregnancy rate | end of 2013 (up to 2 years)

SECONDARY OUTCOMES:
live birth rate | end of 2013 (up to 2 years)

CONTACTS AND LOCATIONS:
Locations (1):
- Christophe Blockeel, Brussels, Belgium

REFERENCES:
- [Derived] Blockeel C, Knez J, Polyzos NP, De Vos M, Camus M, Tournaye H. Should an intrauterine insemination with donor semen be performed 1 or 2 days after the spontaneous LH rise? A prospective RCT. Hum Reprod. 2014 Apr;29(4):697-703. doi: 10.1093/humrep/deu022. Epub 2014 Feb 18. PMID 24549212